CLINICAL TRIAL: NCT05349656
Title: Comparing the Postoperative Analgesic Efficiency of Trans-muscular Quadratus Lumborum Block Versus PENG Block for Hip Surgery in Pediatrics: A Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of Quadratus Lumborum Block Versus Pericapsular Nerve Group Block in Pediatric Hip Surgery
Acronym: TQL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Hisham mohamed gamal eldine hassan, Principal Investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB NO: 00012098 SN: 0305475
Record Dates: First submitted 2022-04-01; First posted 2022-04-27 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2022-05

CONDITIONS: Pain, Postoperative; Developmental Dislocation of Hip
Keywords: quadratus lumborum block; pericapsular nerve group block; developmental dysplasia of the hip; postoperative analgesia; pediatric; hip surgery
MeSH Terms: conditions — Pain, Postoperative; Hip Dislocation; Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trans muscular quadratus lumborum (TQL) block (Experimental): after induction of general anesthesia (GA), the participant will be placed in the lateral position, and a high-frequency linear ultrasound probe (5-13 MHz) will be placed on the anterior iliac crest. The Petit's triangle (formed of the iliac crest inferiorly and the borders of external abdominal oblique anteriorly and latissimus dorsi (LD) posteriorly) will be identified and then Tracing dorsally from Petit's triangle, the external oblique, and the internal oblique are seen disappearing into an aponeurosis as the quadratus lumborum (QL) appears beneath the LD (anteriorly), and going farther dorsally, the QL, erector spinae, and psoas major (PM) muscles around the transverse process of lumbar vertebra L4 are seen. A 22-gauge needle will be inserted using an in-plane technique along the posterior edge of the probe in the anteromedial direction. The needle tip will be placed between the QL muscle and the PM muscle, then 0.5 ml/kg of 0.25% bupivacaine will be injected.
  Interventions: Procedure: TQL block
- Pericapsular nerve group (PENG) block (Experimental): After induction of GA, the participant will be in the supine position. A linear high-frequency ultrasound probe (5-13MHz) will be initially placed in a transverse plane over the anterior inferior iliac spine (AIIS) and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees; In this view, the ilio-pubic eminence (IPE), the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will be observed. A 22-gauge, 80-mm needle Will be inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, the local anesthetic solution of 0.25% bupivacaine will be injected in 5-mL increments while observing for an adequate fluid spread in this plane for a total volume of 0.5 ml/kg.
  Interventions: Procedure: PENG block

INTERVENTIONS:
Procedure: TQL block — Ultrasonography-guided quadratus lumborum block (QLB) where we will infiltrate local anesthetic solution adjacent to the anterolateral aspect of the quadratus lumborum muscle
  Other Names: transmuscular quadratus lumborum block
  Arms: trans muscular quadratus lumborum (TQL) block
Procedure: PENG block — Ultrasound-guided local anesthetic infiltration will be injected in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly
  Other Names: pericapsular nerve group block
  Arms: Pericapsular nerve group (PENG) block

SUMMARY:
Surgical procedure including hip joint surgery is extremely painful and associated with considerable postoperative pain in children despite the use of systemic opioids.

Caudal block is a common method used for perioperative pain relief in pediatric lower limb surgeries but carries some complications.

Some novel techniques of regional anesthesia were explored including the quadratus lumborum block (QLB), lumbar plexus block, and recently Pericapsular nerve group (PENG) block.

The objective of the current trial is primarily to assess the analgesic efficacy of ultrasound-guided trans-muscular QLB versus ultrasound-guided PENG block in pediatric patients undergoing open hip surgery for developmental dysplasia of the hip (DDH)

DETAILED DESCRIPTION:
During the pre-anesthesia check-up visit, the proposed intervention will be discussed with the eligible participant's parents or caregivers including data about the aim, the advantages, and the expected side effects, and then detailed informed consent will be obtained before recruitment and randomization.

All participants will be premedicated with 0.5mg/kg oral midazolam about 30min before being admitted to the operating room. The routine standard monitoring including electrocardiography (ECG), non-invasive blood pressure (NIBP, oxygen saturation (SpO2), temperature probe, and end-tidal CO2 (EtCO2) will be applied to all participants. Induction of anesthesia will be performed using a face mask with sevoflurane inhalation in oxygen starting with 2% up to 8% till complete loss of consciousness after that peripheral intravenous (IV) line will be secured where fentanyl 1 μg/kg and followed by cisatracurium 0.15mg/kg to facilitate orotracheal intubation. Anesthesia will be maintained by using isoflurane 1.2-1.5% in oxygen air mixture 50%:50% in addition to incremental cisatracurium 0.03mg/kg.

After induction of general anesthesia, the eligible participants will be randomly assigned to one of two equal groups using an allocation sequence which will be generated using permuted block randomization technique and the block size will be variable.

In both interventional groups of participants, the assigned block will be performed after induction of general anesthesia by the same investigator who will have no further role in the study. Surgery will be started about 15 minutes after performing the block.

Fentanyl 1μg/ kg will be administrated in the case of inadequate analgesia which is defined as an increase of heart rate (HR) and/or mean arterial blood pressure (MAP) more than 20% above the pre-operative values. At the end of the surgery, isoflurane will be switched off and extubation will be done after reversal of muscle relaxant with neostigmine 0.05 mg/kg and atropine 0.02 mg/kg where the participants will be transferred to the Post-Anesthesia Care Unit (PACU). Paracetamol (15 mg/kg) will be administered IV every 6 hours in all patients. Postoperative pain will be assessed by FLACC score (Face, leg, activity, cry, consolability). Morphine 0.1 mg /kg IV will be given as rescue analgesia if the FLACC score will be > 3. Postoperative HR and MAP will be recorded postoperatively at 2 h, 4, 8, 12, 24, and 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* American society association (ASA) physical status class I - II.
* Participants who will be scheduled for an elective unilateral open hip surgery for correction of DDH under general anesthesia

Exclusion Criteria:

* Participants with respiratory disease, renal or hepatic insufficiency.
* Infection of the skin in the puncture area.
* Coagulopathy.
* Allergy against any of the drugs to be used (bupivacaine).
* Neuromuscular disease.
* Obesity (body mass index, BMI >30).
* Previous hip surgery.
* Previous analgesic medication, chronic pain.
* Previously known neurological pathologies or central nervous system disorders

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
the time until the first rescue analgesic requirement postoperatively | During the first postoperative 48 hours
  Postoperative pain will be assessed by Face, leg, activity, cry, consolability (FLACC) score at different time points with a minimum score of zero (relaxed & comfortable) to a maximum of 10 (severe discomfort & pain). This will be done by the attending physician either in the PACU or in the ward. If FLACC will come > 3, morphine 0.1 mg/kg will be given as rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed I Elnaggar, MD, Study Director — University of Alexandria
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gurkan Y, Aksu C, Kus A, Toker K, Solak M. One operator's experience of ultrasound guided lumbar plexus block for paediatric hip surgery. J Clin Monit Comput. 2017 Apr;31(2):331-336. doi: 10.1007/s10877-016-9869-x. Epub 2016 Mar 31. PMID 27033707
- [Result] Andreae MH, Andreae DA. Regional anaesthesia to prevent chronic pain after surgery: a Cochrane systematic review and meta-analysis. Br J Anaesth. 2013 Nov;111(5):711-20. doi: 10.1093/bja/aet213. Epub 2013 Jun 28. PMID 23811426
- [Result] Kao SC, Lin CS. Caudal Epidural Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:9217145. doi: 10.1155/2017/9217145. Epub 2017 Feb 26. PMID 28337460
- [Result] Auroy Y, Benhamou D, Bargues L, Ecoffey C, Falissard B, Mercier FJ, Bouaziz H, Samii K. Major complications of regional anesthesia in France: The SOS Regional Anesthesia Hotline Service. Anesthesiology. 2002 Nov;97(5):1274-80. doi: 10.1097/00000542-200211000-00034. PMID 12411815
- [Result] Huang C, Zhang X, Dong C, Lian C, Li J, Yu L. Postoperative analgesic effects of the quadratus lumborum block III and transversalis fascia plane block in paediatric patients with developmental dysplasia of the hip undergoing open reduction surgeries: a double-blinded randomised controlled trial. BMJ Open. 2021 Feb 4;11(2):e038992. doi: 10.1136/bmjopen-2020-038992. PMID 33542037
- [Result] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Result] Aksu C, Cesur S, Kus A. Pericapsular nerve group (PENG) block for postoperative analgesia after open reduction of pediatric congenital dysplasia of the hip. J Clin Anesth. 2020 May;61:109675. doi: 10.1016/j.jclinane.2019.109675. Epub 2019 Dec 1. No abstract available. PMID 31796372
- [Result] Orozco S, Munoz D, Jaramillo S, Herrera AM. Pediatric use of Pericapsular Nerve Group (PENG) block for hip surgical procedures. J Clin Anesth. 2019 Nov;57:143-144. doi: 10.1016/j.jclinane.2019.04.010. Epub 2019 Apr 22. No abstract available. PMID 31022606
- [Result] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Result] Sauter AR. The "Shamrock Method"-a new and promising technique for ultrasound guided lumbar plexus blocks. BJA: British Journal of Anaesthesia. 2013; 111(eLetters Supplement).
- [Result] Sato M, Hara M, Uchida O. An antero-lateral approach to ultrasound-guided lumbar plexus block in supine position combined with quadratus lumborum block using single-needle insertion for pediatric hip surgery. Paediatr Anaesth. 2017 Oct;27(10):1064-1065. doi: 10.1111/pan.13208. No abstract available. PMID 28888083
- [Result] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Result] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Result] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343